CLINICAL TRIAL: NCT02202746
Title: A Phase 2, Open-label, Multicenter, Safety and Efficacy Study of Oral Lucitanib in Patients With FGF Aberrant Metastatic Breast Cancer
Brief Title: A Study to Assess the Safety and Efficacy of the VEGFR-FGFR-PDGFR Inhibitor, Lucitanib, Given to Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to end monotherapy development of the compound in breast cancer.
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-3810-025
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; MBC; HER2 Positive; HER2; Estrogen Receptor Positive; ER; Triple Negative
Keywords: Breast cancer; Metastatic breast cancer; MBC; HER2 positive; HER2+; Estrogen receptor positive; ER+; Triple negative; FGFR1; 11q; FGF aberrant; Biomarker negative; FGF non-aberrant
MeSH Terms: conditions — Breast Neoplasms | interventions — E-3810

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: Lucitanib (CO-3810) 10 mg daily (Experimental): 10 mg of lucitanib daily in patients with FGFR1-amplified or 11q-amplified metastatic breast cancer.
  Interventions: Drug: Lucitanib
- Cohort B: Lucitanib (CO-3810) 15 mg daily (Experimental): 15 mg of lucitanib daily in patients with FGFR1-amplified and 11q-amplified metastatic breast cancer.
  Interventions: Drug: Lucitanib
- Cohort C: Lucitanib (CO-3810) 10 mg daily (Experimental): 10 mg of lucitanib daily in patients with FGFR1 non-amplified and 11q non-amplified metastatic breast cancer.
  Interventions: Drug: Lucitanib

INTERVENTIONS:
Drug: Lucitanib — Lucitanib is a potent, orally available selective inhibitor of the tyrosine kinase activity of fibroblast growth factor receptors (FGFR1-3), vascular endothelial growth factor receptors (VEGFR1-3), and platelet-derived growth factor receptors alpha and beta (PDGFR alpha and beta)
  Other Names: CO-3810

SUMMARY:
The purpose of this study is to determine whether lucitanib is safe and effective in the treatment of patients with FGF aberrant metastatic breast cancer, as well as in the treatment of patients with biomarker negative (FGF non-aberrant) metastatic breast cancer.

DETAILED DESCRIPTION:
Lucitanib is a selective, orally available tyrosine kinase inhibitor targeting FGFR1-3, VEGFR1-3, and PDGFRα and β, with activity in relevant cell lines and animal models.

The first in human trial of lucitanib demonstrated that daily dosing with lucitanib can provide durable clinical responses in patients with FGFR1- or 11q (FGF3, FGF4, Cyclin D1, or FGF19)-amplified breast cancer. RECIST partial responses (PRs) were also observed in patients not known to have FGF abnormalities.

Based on these results, this study is designed to explore the safety and anti-tumor activity of daily lucitanib in breast cancer patients with and without alterations of the FGF pathway.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast cancer relapsed or refractory to approved standard available treatment
* Prior treatment with standard first line therapy in the metastatic setting
* Availability of tumor tissue sufficient for confirmatory testing of FGFR1 and 11q amplification status
* Demonstrated progression of disease by radiological or clinical assessment (Measurable disease according to RECIST Version 1.1 is NOT required for enrollment)
* Estimated life expectancy >6 months

Exclusion Criteria:

* Current or recent treatment with biologic anticancer therapies
* Ongoing AEs from prior anticancer therapies
* Active central nervous system (CNS) metastases
* Clinically significant or uncontrolled hypertension or cardiac disease
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Arizona Oncology Associates, Sedona, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Saint Jude Heritage Medical Center, Fullerton, California
  - Moores UCSD Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - University of California San Francisco, San Francisco, California
  - Central Coast Medical Oncology Group, Santa Maria, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Deerfield Beach, Florida
  - Memorial West Cancer Center, Hollywood, Florida
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Cooper University Hospital, Voorhees Township, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Breast Center, New York, New York
  - Sciode Medical Associates, PLLC, The Bronx, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Austin Central, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - US Oncology, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Derived] Liao M, Zhou J, Wride K, Lepley D, Cameron T, Sale M, Xiao J. Population Pharmacokinetic Modeling of Lucitanib in Patients with Advanced Cancer. Eur J Drug Metab Pharmacokinet. 2022 Sep;47(5):711-723. doi: 10.1007/s13318-022-00773-w. Epub 2022 Jul 18. PMID 35844029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 178 patients were recruited from 32 sites in the United States.
Groups:
- Lucitanib (CO-3810) 10 mg QD: 10 mg of lucitanib daily in continuous 28-day treatment cycles until tumor progression, unacceptable toxicity, or withdrawal for other reasons
- Lucitanib (CO-3810) 15 mg QD: 15 mg of lucitanib daily in continuous 28-day treatment cycles until tumor progression, unacceptable toxicity, or withdrawal for other reasons
Period: Overall Study
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Started | 109 | 69
Completed | 109 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD | Total
Number analyzed (Participants) | 109 | 69 | 178
Age, Continuous [Median (Full Range); unit: years] | 57.0 [27 to 82] | 53.0 [27 to 80] | 55.0 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 67 | 176
  Male | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 61 | 148
  Asian | 5 | 3 | 8
  Black | 10 | 1 | 11
  Not provided | 4 | 3 | 7
  Unknown/Not assessed | 2 | 1 | 3
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 97 | 61 | 158
  Not Provided | 4 | 2 | 6
Number of Prior Anticancer Therapies [Median (Full Range); unit: Therapies] | 6.0 [1 to 18] | 6.0 [1 to 16] | 6.0 [1 to 18]
Fibroblast Growth Factor (FGF) Status [Count of Participants; unit: Participants] — FGFR1 and 11q are genes that are amplified in a percentage of breast cancers. Sites were required to submit archival tumor specimens for all enrolled patients for central laboratory confirmation of FGFR1 or 11q amplification status. Patients were categorized based on results indicating FGFR1 amplification, 11q amplification, both FGFR1 and 11q amplification, or non-amplification of either gene (negative).
  Participants
    11q | 34 | 25 | 59
    FGFR1 | 50 | 28 | 78
    FGFR1 & 11q | 18 | 10 | 28
    Negative | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 as Determined by the Investigator
Description: The primary efficacy endpoint of PFS was calculated as 1+ the number of days from the date of first dose of study drug to disease progression or death due to any cause, whichever occurs first. Patients without a documented event of progression were censored on the date of their last adequate tumor assessment (i.e., radiologic assessment), or the date of randomization if no tumor assessments were performed. Progression events were determined by the investigator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 29 months
Population: Efficacy population: all patients who have received at least one dose of lucitanib and are confirmed as FGR1-, 11q-amplified, or FGF non-amplified per the central laboratory
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 107 | 67
Days | 93 [78 to 140] | 77 [50 to 86]

2. Secondary Outcome: Objective Response Rate (ORR) by RECIST v1.1
Description: ORR is the percentage of patients with a best response of CR or PR according to RECIST v1.1. The best response is recorded from the start of the treatment (Day 1) until disease progression or recurrence. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 29 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- All Patients: The total efficacy population analyzed for response
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD | All Patients
Number analyzed (Participants) | 106 | 67 | 173
percentage of participants | 4.7 | 1.5 | 3.5

3. Secondary Outcome: Duration of Response (DR) by RECIST v1.1
Description: DR for complete response (CR) and partial response (PR) was measured from the date that any of these best confirmed responses was first recorded until the first date that PD was objectively documented. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 29 months
Population: Efficacy population for patients who had a confirmed CR or PR
Measure: Median (Full Range); unit: Days
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 5 | 1
Days | 175 [44 to 209] | 336 [336 to 336]

4. Secondary Outcome: Disease Control Rate (DCR) by RECIST v1.1
Description: The DCR is defined as the percentage of patients with a best response rate of CR, PR, or SD for at least 12 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 29 months
Population: Efficacy population only
Measure: Number; unit: percentage of patients
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD | All Patients
Number analyzed (Participants) | 106 | 67 | 173
percentage of patients | 48.1 | 34.3 | 42.8

5. Secondary Outcome: Comparative Pharmacokinetics (PK) of the Lucitanib Capsule Formulation vs. Tablet Formulation - Cmax
Description: The comparative PK study was a within-patient comparison of tablet and capsule formulations of lucitanib administered orally. PK sampling was performed at specified time points on each of the following two days: • Day -7: patients received a single administration of 10 mg or 15 mg lucitanib tablet formulation • Day 1: patients received a single administration of 10 mg or 15 mg lucitanib in capsule formulation. Cmax = maximum concentration following administration of lucitanib.
Time Frame: Study Day -7 to Study Day 1, or approximately 8 days
Population: PK parameters were assessed in a subset of patients (N=15)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lucitanib (CO-3810) 10 mg QD: 10 mg of lucitanib tablet or capsule given orally
- Lucitanib (CO-3810) 15 mg QD: 15 mg of lucitanib tablet or capsule given orally
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 9 | 6
ng/mL
  Tablet | 292 (156) | 278 (99.8)
  Capsule | 265 (137) | 285 (121)

6. Secondary Outcome: Comparative Pharmacokinetics (PK) of the Lucitanib Capsule Formulation vs. Tablet Formulation - Tmax
Description: The comparative PK study was a within-patient comparison of tablet and capsule formulations of lucitanib administered orally. PK sampling was performed at specified time points on each of the following two days: • Day -7: patients received a single administration of 10 mg or 15 mg lucitanib tablet formulation • Day 1: patients received a single administration of 10 mg or 15 mg lucitanib in capsule formulation. Tmax = time to maximum concentration following administration of lucitanib
Time Frame: Study Day -7 to Study Day 1, or approximately 8 days
Population: PK parameters were assessed in a subset of patients (N=15)
Measure: Median (Full Range); unit: Hours
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 9 | 6
Hours
  Tablet | 1.0 [0.5 to 4.0] | 1.0 [0.5 to 2.5]
  Capsule | 1.5 [1.0 to 4.0] | 1.0 [1.0 to 2.5]

7. Secondary Outcome: Comparative Pharmacokinetics (PK) of the Lucitanib Capsule Formulation vs. Tablet Formulation - AUClast
Description: The comparative PK study was a within-patient comparison of tablet and capsule formulations of lucitanib administered orally. PK sampling was performed at specified time points on each of the following two days: • Day -7: patients received a single administration of 10 mg or 15 mg lucitanib tablet formulation • Day 1: patients received a single administration of 10 mg or 15 mg lucitanib in capsule formulation. AUClast = area under the plasma concentration time curve from time 0 to the last quantifiable time point (24 hour)
Time Frame: Study Day -7 to Study Day 1, or approximately 8 days
Population: PK parameters were assessed in a subset of patients (N=15)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 9 | 6
h*ng/mL
  Tablet | 2550 (1150) | 2840 (1230)
  Capsule | 2650 (1380) | 2420 (613)

8. Secondary Outcome: Comparative Pharmacokinetics (PK) of the Lucitanib Capsule Formulation vs. Tablet Formulation - AUCinf
Description: The comparative PK study was a within-patient comparison of tablet and capsule formulations of lucitanib administered orally. PK sampling was performed at specified time points on each of the following two days: • Day -7: patients received a single administration of 10 mg or 15 mg lucitanib tablet formulation • Day 1: patients received a single administration of 10 mg or 15 mg lucitanib in capsule formulation. AUCinf = area under the plasma concentration time curve from 0 to infinity
Time Frame: Study Day -7 to Study Day 1, or approximately 8 days
Population: PK parameters were assessed in a subset of patients (N=15)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 9 | 6
h*ng/mL
  Tablet | 4780 (2140) | 5720 (3760)
  Capsule | 5680 (2730) | 4620 (1620)

9. Secondary Outcome: Relative Bioavailability Analysis for Tablet vs Capsule - Cmax, AUClast, AUCinf
Description: Relative bioavailability of lucitanib was evaluated by comparison of (log-transformed) AUClast, Cmax and AUCinf of the tablet formulation to the capsule formulation using an analysis of variance (ANOVA) model with treatment as a fixed effect. The geometric means, ratio of the geometric means and 90% confidence intervals (CI) on the ratio of Tablet to Capsule (T:R) were presented for AUClast, Cmax and AUCinf. The CIs on the ratio of untransformed PK parameters were derived through reverse transformation of the 90% CI of the difference in the log scale to the 90% CI of the ratio in the original scale.
Time Frame: Study Day -7 to Study Day 1, or approximately 8 days
Population: PK parameters were assessed in a subset of patients (N=15).
Measure: Number (90% Confidence Interval); unit: Percentage (tablet/capsule)
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
Number analyzed (Participants) | 9 | 6
Percentage (tablet/capsule)
  Cmax Geometric Mean Ratio | 111.73 [70.35 to 177.45] | 100.56 [64.59 to 156.55]
  AUClast Geometric Mean Ratio | 97.58 [60.61 to 157.09] | 112.2 [78.73 to 159.89]
  AUCinf Geometric Mean Ratio | 82.9 [51.75 to 132.81] | 114.23 [70.09 to 186.15]

10. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the number of days from the date of first dose of study drug to the date of death (due to any cause). Patients without a known date of death will be censored on the date the patient was last known to be alive.
Time Frame: Cycle 1 Day 1 to date of death, assessed up to 29 months
Population: Intent to treat population by initial treatment and overall
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD | All Patients
Number analyzed (Participants) | 109 | 69 | 178
Months | 15.0 [10.7 to 17.3] | 7.7 [6.1 to 10.3] | 10.7 [8.5 to 13.7]

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) Total Score
Description: FACT-B is used for assessment of health-related quality of life (QoL) in participants with breast cancer. It consists of 37 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and breast cancer subscale (10 items) ranging from 0 to 40; high subscale score represents a better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. FACT-B Total Score is derived from adding the five subscale scores. Total possible score ranges from 0 to 148. High scale score represents a better QoL.
Time Frame: From Cycle 1 Day 1 until end of treatment, assessed up to 29 months
Population: Efficacy Population defined as all patients who have received at least one dose of Lucitanib and have at least one post-baseline Investigator Overall Objective Tumor Assessment. 'Overall Number of Participants Analyzed'=participants who completed both a baseline FACT-B assessment and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD | All Patients
Number analyzed (Participants) | 80 | 46 | 126
units on a scale | -2.422 (15.5134) | -7.586 (17.0709) | -4.307 (16.2248)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of first dose of lucitanib through 28 days after last dose protocol-specified treatment administration, up to approximately 30 months. In addition, study procedure-related AEs that occur after signing of the informed consent form and before administration of lucitanib were also collected.
Description: If a patient experiences the same preferred term (system organ class) multiple times, then the patient will be counted only once for that preferred term (system organ class).
Arm/Group | Lucitanib (CO-3810) 10 mg QD | Lucitanib (CO-3810) 15 mg QD
All-Cause Mortality (participants affected / at risk) | 5/109 | 7/69
Serious Adverse Events (participants affected / at risk) | 31/109 | 22/69
Other Adverse Events (participants affected / at risk) | 107/109 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucitanib (CO-3810) 10 mg QD (N=109) | Lucitanib (CO-3810) 15 mg QD (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Ammonia increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lucitanib (CO-3810) 10 mg QD (N=109) | Lucitanib (CO-3810) 15 mg QD (N=69)
Anaemia (Blood and lymphatic system disorders) | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 9
Hypothyroidism (Endocrine disorders) | 41 | 34
Vision blurred (Eye disorders) | 7 | 3
Abdominal distension (Gastrointestinal disorders) | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 16 | 9
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 20 | 12
Diarrhoea (Gastrointestinal disorders) | 33 | 19
Dry mouth (Gastrointestinal disorders) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 10 | 4
Nausea (Gastrointestinal disorders) | 53 | 33
Vomiting (Gastrointestinal disorders) | 35 | 24
Fatigue (General disorders) | 55 | 37
Mucosal inflammation (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 13 | 4
Pain (General disorders) | 7 | 3
Pyrexia (General disorders) | 8 | 2
Sinusitis (Infections and infestations) | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 14 | 10
Alanine aminotransferase increased (Investigations) | 9 | 4
Aspartate aminotransferase increased (Investigations) | 10 | 4
Blood alkaline phosphatase increased (Investigations) | 9 | 3
Blood bilirubin increased (Investigations) | 6 | 4
Blood thyroid stimulating hormone increased (Investigations) | 6 | 2
Ejection fraction decreased (Investigations) | 3 | 5
Platelet count decreased (Investigations) | 4 | 6
Weight decreased (Investigations) | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 36 | 21
Dehydration (Metabolism and nutrition disorders) | 8 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Dizziness (Nervous system disorders) | 15 | 5
Dysgeusia (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 42 | 24
Anxiety (Psychiatric disorders) | 7 | 6
Depression (Psychiatric disorders) | 8 | 7
Insomnia (Psychiatric disorders) | 11 | 6
Haematuria (Renal and urinary disorders) | 3 | 6
Proteinuria (Renal and urinary disorders) | 22 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 5 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Hot flush (Vascular disorders) | 5 | 4
Hypertension (Vascular disorders) | 85 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All parties agree to submit all manuscripts or abstracts to all other parties 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties. The sponsor may request a delay in publication if there are important intellectual property concerns relating to publication, but does not have the right to suppress publication of the study results indefinitely.

DOCUMENTS (2):
  • Study Protocol (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02202746/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02202746/SAP_001.pdf